CLINICAL TRIAL: NCT01473381
Title: A Double-blind, Placebo- and Active-controlled, Fixed-dose Study of Vilazodone in Patients With Major Depressive Disorder
Brief Title: Safety and Efficacy of Vilazodone in Major Depressive Disorder
Acronym: VLZ-MD-01
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VLZ-MD-01
Record Dates: First submitted 2011-11-14; First posted 2011-11-17 (Estimated); Results first posted 2014-08-08 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Vilazodone Hydrochloride; Citalopram

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Participants received 2 placebo to vilazodone tablets, and 1 placebo to citalopram capsule orally once daily for the 11 weeks of the study.
  Interventions: Drug: Placebo to citalopram; Drug: Placebo to vilazodone
- Vilazodone 20 mg/day (Experimental): Participants received 1 vilazodone tablet, 1 placebo to vilazodone tablet, and 1 placebo to citalopram capsule orally once daily for the 11 weeks of the study. Participants received vilazodone 10 mg/day during Week 1, vilazodone 20 mg/day during Weeks 2 to 10, and vilazodone 10 mg/day during Week 11.
  Interventions: Drug: Vilazodone; Drug: Placebo to citalopram; Drug: Placebo to vilazodone
- Vilazodone 40 mg/day (Experimental): Participants received 1 placebo to vilazodone tablet, 1 vilazodone tablet, and 1 placebo to citalopram capsule orally once daily during Weeks 1 and 2 of the study. Participants received 2 vilazodone tablets and 1 placebo to citalopram capsule orally once daily during Weeks 3 -10 of the study. Participants received vilazodone 10 mg/day during Week 1, vilazodone 20/day mg during Week 2, and vilazodone 40 mg/day during Weeks 3 to 10. During Week 11, participants received vilazodone 20 mg/day for 4 days and 10 mg/day for 3 days.
  Interventions: Drug: Vilazodone; Drug: Placebo to citalopram; Drug: Placebo to vilazodone
- Citalopram 40 mg/day (Active Comparator): Participants received 2 placebo vilazodone tablets, and 1 citalopram capsule once daily for the 11 weeks of the study. Participants received citalopram 20 mg/day during Weeks 1 and 2, citalopram 40 mg/day during Weeks 3 to 10, and citalopram 20 mg/day during Week 11.
  Interventions: Drug: Placebo to vilazodone; Drug: Citalopram

INTERVENTIONS:
Drug: Vilazodone — Vilazodone was supplied as film-coated tablets.
  Other Names: Viibryd
  Arms: Vilazodone 20 mg/day; Vilazodone 40 mg/day
Drug: Placebo to citalopram — Placebo to citalopram was supplied as a capsule.
  Other Names: Celexa
  Arms: Placebo; Vilazodone 20 mg/day; Vilazodone 40 mg/day
Drug: Placebo to vilazodone — Placebo to vilazodone was supplied as film-coated tablets.
Drug: Citalopram — Citalopram was supplied as encapsulated tablets.
  Other Names: Celexa
  Arms: Citalopram 40 mg/day

SUMMARY:
The purpose of this study was to evaluate the efficacy, safety, and tolerability of 2 fixed dose levels of vilazodone compared to placebo in patients with major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18-70 years of age.
* Currently meet the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria for Major Depressive Disorder.
* The patient's current major depressive episode must be at least 8 weeks and no longer than 12 months in duration.

Exclusion Criteria:

* Women who are pregnant, women who will be breastfeeding during the study, and women of childbearing potential who are not practicing a reliable method of birth control.
* Patients with a history of meeting DSM-IV-TR criteria for:

  * Any manic, hypomanic or mixed episode, including bipolar disorder and substance-induced manic, hypomanic, or mixed episode
  * Any depressive episode with psychotic or catatonic features
  * Panic disorder with or without agoraphobia
  * Obsessive-compulsive disorder
  * Schizophrenia, schizoaffective, or other psychotic disorder
  * Bulimia or anorexia nervosa
  * Presence of borderline personality disorder or antisocial personality disorder
  * Mental retardation, dementia, amnesia, or other cognitive disorders.
* Patients who are considered a suicide risk.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1162 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Gommoll, MS, Study Director — Forest Laboratories
Locations (54):
- United States (54):
  - Forest Investigative Site 036, Birmingham, Alabama
  - Forest Investigative Site 016, Dothan, Alabama
  - Forest Investigative Site 033, Scottsdale, Arizona
  - Forest Investigative Site 027, Fayetteville, Arkansas
  - Forest Investigative Site 029, Cerritos, California
  - Forest Investigative Site 002, Costa Mesa, California
  - Forest Investigative Site 019, Murrieta, California
  - Forest Investigative Site 025, Oceanside, California
  - Forest Investigative Site 043, Orange, California
  - Forest Investigative Site 003, Redlands, California
  - Forest Investigative Site 046, Sherman Oaks, California
  - Forest Investigative Site 057, Upland, California
  - Forest Investigative Site 034, Cromwell, Connecticut
  - Forest Investigative Site 038, Fort Myers, Florida
  - Forest Investigative Site 018, Gainsville, Florida
  - Forest Investigative Site 055, Hallandale, Florida
  - Forest Investigative Site 063, Jacksonville, Florida
  - Forest Investigative Site 035, Miami, Florida
  - Forest Investigative Site 030, Orlando, Florida
  - Forest Investigative Site 062, Orlando, Florida
  - Forest Investigative Site 045, Pembroke Pines, Florida
  - Forest Investigative Site 051, Tampa, Florida
  - Forest Investigative Site 032, West Palm Beach, Florida
  - Forest Investigative Site 022, Winter Park, Florida
  - Forest Investigative Site 060, Atlanta, Georgia
  - Forest Investigative Site 037, Chicago, Illinois
  - Forest Investigative Site 050, Chicago, Illinois
  - Forest Investigative Site 040, Indianapolis, Indiana
  - Forest Investigative Site 012, Lafayette, Indiana
  - Forest Investigative Site 053, Prairie Village, Kansas
  - Forest Investigative Site 020, Baltimore, Maryland
  - Forest Investigative Site 031, Boston, Massachusetts
  - Forest Investigative Site 061, Las Vegas, Nevada
  - Forest Investigative Site 024, Willingboro, New Jersey
  - Forest Investigative Site 010, Albuquerque, New Mexico
  - Forest Investigative Site 011, Albuquerque, New Mexico
  - Forest Investigative Site 004, Brooklyn, New York
  - Forest Investigative Site 007, Cedarhurst, New York
  - Forest Investigative Site 058, New York, New York
  - Forest Investigative Site 047, New York, New York
  - Forest Investigative Site 039, Cincinnati, Ohio
  - Forest Investigative Site 042, Oklahoma City, Oklahoma
  - Forest Investigative Site 048, Oklahoma City, Oklahoma
  - Forest Investigative Site 066, Portland, Oregon
  - Forest Investigative Site 014, Allentown, Pennsylvania
  - Forest Investigative Site 049, Bridgeville, Pennsylvania
  - Forest Investigative Site 064, Memphis, Tennessee
  - Forest Investigative Site 013, Austin, Texas
  - Forest Investigative Site 021, Dallas, Texas
  - Forest Investigative Site 059, Bellevue, Washington
  - Forest Investigative Site 065, Seattle, Washington
  - Forest Investigative Site 054, Spokane, Washington
  - Forest Investigative Site 052, Middleton, Wisconsin
  - Forest Investigative Site 056, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Kornstein S, Chang CT, Gommoll CP, Edwards J. Vilazodone efficacy in subgroups of patients with major depressive disorder: a post-hoc analysis of four randomized, double-blind, placebo-controlled trials. Int Clin Psychopharmacol. 2018 Jul;33(4):217-223. doi: 10.1097/YIC.0000000000000217. PMID 29608461
- [Derived] Rele S, Millet R, Kim S, Paik JW, Kim S, Masand PS, Patkar AA. An 8-Week Randomized, Double-Blind Trial Comparing Efficacy, Safety, and Tolerability of 3 Vilazodone Dose-Initiation Strategies Following Switch From SSRIs and SNRIs in Major Depressive Disorder. Prim Care Companion CNS Disord. 2015 Aug 6;17(4):10.4088/PCC.14m01734. doi: 10.4088/PCC.14m01734. eCollection 2015. PMID 26693034
- [Derived] Clayton AH, Gommoll C, Chen D, Nunez R, Mathews M. Sexual dysfunction during treatment of major depressive disorder with vilazodone, citalopram, or placebo: results from a phase IV clinical trial. Int Clin Psychopharmacol. 2015 Jul;30(4):216-23. doi: 10.1097/YIC.0000000000000075. PMID 26039688
- [Derived] Mathews M, Gommoll C, Chen D, Nunez R, Khan A. Efficacy and safety of vilazodone 20 and 40 mg in major depressive disorder: a randomized, double-blind, placebo-controlled trial. Int Clin Psychopharmacol. 2015 Mar;30(2):67-74. doi: 10.1097/YIC.0000000000000057. PMID 25500685

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Vilazodone 20 mg/Day | Vilazodone 40 mg/Day | Citalopram 40 mg/Day
Started | 290 | 292 | 291 | 289
Safety Population | 281 | 288 | 287 | 282
Completed | 210 | 199 | 189 | 200
Not Completed | 80 | 93 | 102 | 89
Not completed — Adverse Event | 8 | 20 | 25 | 17
Not completed — Insufficient Therapeutic Response | 10 | 1 | 2 | 3
Not completed — Protocol Violation | 17 | 23 | 19 | 17
Not completed — Withdrawal of Consent | 20 | 21 | 20 | 26
Not completed — Lost to Follow-up | 25 | 28 | 35 | 23
Not completed — Other Reasons | 0 | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Safety population: All randomized participants who received at least 1 dose of double-blind investigational product (placebo, vilazodone, or citalopram).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vilazodone 20 mg/Day | Vilazodone 40 mg/Day | Citalopram 40 mg/Day | Total
Number analyzed (Participants) | 281 | 288 | 287 | 282 | 1138
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (13.0) | 41.7 (12.7) | 40.8 (13.2) | 42.6 (12.6) | 41.8 (12.8)
Age, Customized [Number; unit: participants]
  < 20 years | 5 | 2 | 9 | 2 | 18
  ≥ 20-29 years | 63 | 62 | 63 | 53 | 241
  ≥ 30-39 years | 48 | 59 | 68 | 59 | 234
  ≥ 40-49 years | 73 | 88 | 62 | 76 | 299
  ≥ 50-59 years | 66 | 50 | 62 | 66 | 244
  ≥ 60 years | 26 | 27 | 23 | 26 | 102
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158 | 166 | 164 | 165 | 653
  Male | 123 | 122 | 123 | 117 | 485
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 59 | 55 | 43 | 53 | 210
  Not Hispanic or Latino | 222 | 233 | 244 | 229 | 928
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 197 | 205 | 202 | 184 | 788
  Black or African American | 71 | 73 | 74 | 83 | 301
  Asian | 7 | 7 | 3 | 3 | 20
  American Indian or Alaska Native | 3 | 0 | 2 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 2 | 1 | 4
  Other | 3 | 2 | 4 | 7 | 16
Weight [Mean (Standard Deviation); unit: kg] | 82.27 (17.02) | 82.55 (18.16) | 82.45 (17.85) | 82.37 (18.30) | 82.41 (17.82)
Weight [Median (Full Range); unit: kg] | 82.50 [46.5 to 127.1] | 82.40 [45.0 to 137.9] | 82.10 [48.8 to 132.9] | 79.50 [46.6 to 151.6] | 81.60 [45.0 to 151.6]
Height [Mean (Standard Deviation); unit: cm] | 169.03 (9.38) | 168.86 (9.72) | 169.87 (9.71) | 169.78 (9.57) | 169.39 (9.60)
Height [Median (Full Range); unit: cm] | 167.60 [144.8 to 198.1] | 167.60 [147.3 to 195.6] | 168.90 [146.0 to 193.0] | 169.00 [144.8 to 200.7] | 168.50 [144.8 to 200.7]
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter squared] | 28.70 (5.40) | 28.79 (5.49) | 28.45 (5.43) | 28.36 (5.17) | 28.58 (5.37)
Body Mass Index (BMI) [Median (Full Range); unit: kilograms per meter squared] | 28.30 [18.5 to 40.0] | 28.20 [18.4 to 39.6] | 27.80 [18.3 to 40.0] | 27.90 [18.0 to 39.9] | 28.10 [18.0 to 40.0]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score at Week 10
Description: The MADRS is a clinician-rated scale based on participant interviews. The scale assesses depressive symptomatology that occurred in participants during the week preceding each interview. Participants were rated on 10 items: Apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Each item was scored on a 7-point scale from 0 (no symptoms) to 6 (symptoms of maximum severity). The total score was the sum of the scores of the 10 items and ranged from 0 to 60. A higher score indicates more depressive symptomatology. A negative change score indicates improvement.
Time Frame: Baseline to Week 10
Population: Intent-to-treat population: All randomized participants who received at least 1 dose of placebo, vilazodone, or citalopram and who had a baseline and at least 1 post-baseline assessment of the MADRS total score.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Vilazodone 20 mg/Day | Vilazodone 40 mg/Day | Citalopram 40 mg/Day
Number analyzed (Participants) | 281 | 288 | 284 | 280
Units on a scale | -14.76 (0.62) | -17.33 (0.63) | -17.58 (0.65) | -17.50 (0.64)
Statistical Analysis 1: Comparison: Placebo vs Vilazodone 20 mg/Day; Test type: Superiority or Other; p = 0.0073, Mixed-effect model — P-value was adjusted for multiplicity; Mean Difference (Final Values) = -2.57, 95% CI 2-sided [-4.30 to -0.84]
Statistical Analysis 2: Comparison: Placebo vs Vilazodone 40 mg/Day; Test type: Superiority or Other; p = 0.0034, Mixed-effect model — P-value was adjusted for multiplicity; Mean Difference (Final Values) = -2.82, 95% CI 2-sided [-4.57 to -1.06]
Statistical Analysis 3: Comparison: Placebo vs Citalopram 40 mg/Day; Test type: Superiority or Other; p = 0.0020, Mixed-effect model — P-value was provided for assay sensitivity. It was not adjusted for multiplicity; Mean Difference (Final Values) = -2.74, 95% CI 2-sided [-4.48 to -1.00]

2. Secondary Outcome: Change From Baseline to Week 10 in the Clinical Global Impressions-Severity (CGI-S) Scale Score
Description: The Clinical Global Impressions-Severity scale is a clinician-rated scale used to rate the severity of the participant's current state of mental illness compared with a patient population with major depressive disorder. In particular, the clinician is asked to respond to the following question: "Considering your total clinical experience with this population, how mentally ill is the patient at this time?" The patient is rated on the following 7-point scale: 1-normal, not at all ill, 2-borderline ill, 3-mildly ill, 4-moderately ill, 5-markedly ill, 6-severely ill, 7-among the most extremely ill patients. A higher score indicates more mental illness. A negative change score indicates improvement.
Time Frame: Baseline to Week 10
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Vilazodone 20 mg/Day | Vilazodone 40 mg/Day | Citalopram 40 mg/Day
Number analyzed (Participants) | 281 | 288 | 284 | 280
Units on a scale | -1.53 (0.08) | -1.88 (0.08) | -1.86 (0.08) | -1.88 (0.08)
Statistical Analysis 1: Comparison: Placebo vs Vilazodone 20 mg/Day; Test type: Superiority or Other; p = 0.0073, Mixed-effect model — P-value was adjusted for multiplicity; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.58 to -0.13]
Statistical Analysis 2: Comparison: Placebo vs Vilazodone 40 mg/Day; Test type: Superiority or Other; p = 0.0097, Mixed-effect model — P-value was adjusted for multiplicity; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-0.55 to -0.10]
Statistical Analysis 3: Comparison: Placebo vs Citalopram 40 mg/Day; Test type: Superiority or Other; p = 0.0025, Mixed-effect model — P-value was provided for assay sensitivity. It was not adjusted for multiplicity; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.57 to -0.12]

3. Secondary Outcome: Percentage of Participants With a Montgomery-Åsberg Depression Rating Scale (MADRS) Sustained Response
Description: The MADRS is a clinician-rated scale based on participant interviews. The scale assesses depressive symptomatology that occurred in participants during the week preceding each interview. Participants were rated on 10 items: Apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Each item was scored on a 7-point scale from 0 (no symptoms) to 6 (symptoms of maximum severity). The total score was the sum of the scores of the 10 items and ranged from 0 to 60. A higher score indicates more depressive symptomatology. A MADRS sustained response was defined as a MADRS total score ≤ 12 for at least the last 2 visits during the double-blind treatment period (Weeks 1-10). A total MADRS score ≤ 12 corresponds to an average score of 1 per item and is indicative of very low level of depressive symptoms.
Time Frame: Baseline to Week 10
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Vilazodone 20 mg/Day | Vilazodone 40 mg/Day | Citalopram 40 mg/Day
Number analyzed (Participants) | 281 | 288 | 284 | 280
Percentage of participants | 26.3 [21.2 to 31.5] | 29.9 [24.6 to 35.1] | 33.5 [28.0 to 38.9] | 31.1 [25.7 to 36.5]
Statistical Analysis 1: Comparison: Placebo vs Vilazodone 20 mg/Day; Test type: Superiority or Other; p = 0.3563, Cochran-Mantel-Haenszel — P-value was adjusted for multiplicity; The Mean Difference (Final Values), as well as 95% Confidence Interval, are in units of percentage; Mean Difference (Final Values) = 3.5, 95% CI 2-sided [-3.9 to 10.9]
Statistical Analysis 2: Comparison: Placebo vs Vilazodone 40 mg/Day; Test type: Superiority or Other; p = 0.1611, Cochran-Mantel-Haenszel — P-value was adjusted for multiplicity; The Mean Difference (Final Values), as well as 95% Confidence Interval, are in units of percentage; Mean Difference (Final Values) = 7.1, 95% CI 2-sided [-0.4 to 14.6]
Statistical Analysis 3: Comparison: Placebo vs Citalopram 40 mg/Day; Test type: Superiority or Other; p = 0.2672, Cochran-Mantel-Haenszel — P-value was provided for assay sensitivity. It was not adjusted for multiplicity; The Mean Difference (Final Values), as well as 95% Confidence Interval, are in units of percentage; Mean Difference (Final Values) = 4.7, 95% CI 2-sided [-2.7 to 12.2]

ADVERSE EVENTS:
Time Frame: From the time that the participant signs the informed consent form until 30 days after the last dose of treatment.
Description: Safety population: All randomized participants who received at least 1 dose of double-blind investigational product (placebo, vilazodone, or citalopram).
Arm/Group | Placebo | Vilazodone 20 mg/Day | Vilazodone 40 mg/Day | Citalopram 40 mg/Day
Serious Adverse Events (participants affected / at risk) | 3/281 | 4/288 | 4/287 | 6/282
Other Adverse Events (participants affected / at risk) | 124/281 | 168/288 | 177/287 | 147/282
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=281) | Vilazodone 20 mg/Day (N=288) | Vilazodone 40 mg/Day (N=287) | Citalopram 40 mg/Day (N=282)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Asthma (Immune system disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bipolar I disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Cardiomegaly (Cardiac disorders) | 0 | 1 | 0 | 0
Diverticulitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Electrocardiogram ST segment abnormal (Investigations) | 1 | 0 | 0 | 0
Gastric disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Hospitalisation (Surgical and medical procedures) | 0 | 0 | 0 | 1
Ilium fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Migraine with aura (Nervous system disorders) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Somnolence (Psychiatric disorders) | 0 | 0 | 1 | 0
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1 | 0
Traumatic renal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wrist fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Abscess Neck (Infections and infestations) | 1 | 0 | 0 | 0
Abscess Oral (Infections and infestations) | 1 | 0 | 0 | 0
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=281) | Vilazodone 20 mg/Day (N=288) | Vilazodone 40 mg/Day (N=287) | Citalopram 40 mg/Day (N=282)
Diarrhoea (Gastrointestinal disorders) | 26 | 75 | 76 | 30
Nausea (Gastrointestinal disorders) | 23 | 62 | 69 | 55
Headache (Nervous system disorders) | 39 | 42 | 41 | 42
Dry mouth (Gastrointestinal disorders) | 14 | 22 | 19 | 18
Vomiting (Gastrointestinal disorders) | 7 | 11 | 19 | 5
Dizziness (Nervous system disorders) | 20 | 18 | 18 | 19
Somnolence (Psychiatric disorders) | 10 | 11 | 18 | 22
Insomnia (Psychiatric disorders) | 8 | 19 | 16 | 12
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 13 | 14 | 15 | 14
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 11 | 12 | 13 | 15
Fatigue (General disorders) | 9 | 11 | 11 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study.

Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.